CLINICAL TRIAL: NCT00000412
Title: Prevention of Osteoporosis After Cardiac Transplantation
Brief Title: Osteoporosis Prevention After Heart Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AR046124 (NIH); R01AR046124 (NIH); NIAMS-008 (Other: NIAMS)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Osteoporosis; Cardiac Transplantation
Keywords: Osteoporosis; Osteopenia; Heart transplant; Bone fracture; Bone density; Dual energy x-ray absorptiometry
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Fractures, Bone | interventions — Alendronate; Calcitriol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group A (Active Comparator): Group A active alendronate (10 mg/day) and placebo calcitriol.
  Interventions: Drug: Alendronate; Drug: Placebo Calcitriol
- Group B (Placebo Comparator): We will give Group B placebo alendronate and active calcitriol (0.25 micrograms BID).
  Interventions: Drug: Calcitriol; Drug: Placebo Alendronate

INTERVENTIONS:
Drug: Alendronate
  Arms: Group A
Drug: Calcitriol
  Arms: Group B
Drug: Placebo Alendronate
  Arms: Group B
Drug: Placebo Calcitriol
  Arms: Group A

SUMMARY:
During the first year after a heart transplant, people often rapidly lose bone from their spine and hips. About 35 percent of people who receive heart transplants will suffer broken bones during the first year after transplantation. This study will compare the safety and effectiveness of the drug alendronate (Fosamax) and the active form of vitamin D (calcitriol) in preventing bone loss at the spine and hip after a heart transplant.

In this study, people who have had a successful heart transplant will receive either active alendronate and a "dummy pill" instead of calcitriol, or active calcitriol and a dummy pill instead of alendronate for the first year after their transplant, starting within 1 month after transplant surgery. We will measure bone density in the hip and spine at the start of the study and after 6 and 12 months, and will also check for broken bones in the spine. This research should lead to ways of preventing this crippling form of osteoporosis.

DETAILED DESCRIPTION:
We will enroll patients who have undergone cardiac transplantation into a randomized, double-blind, 12-month study of the efficacy and safety of calcitriol (Rocaltrol) and alendronate sodium (Fosamax) in the prevention of bone loss after transplantation. We will give all participants standard pre- and post-transplantation management and immunosuppressive therapy, three tablets of calcium citrate (Citracal + D, each containing 315 mg of elemental calcium and 200 IU of vitamin D), and a multivitamin providing 400 units of vitamin D daily. We will randomize participants to one of two active treatment groups within 1 month of transplantation. We will give Group A active alendronate (10 mg/day) and placebo calcitriol. We will give Group B placebo alendronate and active calcitriol (0.25 micrograms BID). The primary efficacy endpoint is the change in spine bone mineral density (BMD) during the first 6 months after transplantation. The secondary efficacy endpoint is the change in hip BMD during the first year after transplantation. We will also monitor the incidence of vertebral fracture.

We will invite eligible subjects to participate in the study. We will offer patients who elect not to participate in the therapeutic trial the opportunity to have serial BMD measurements at the same intervals as treated subjects and to be followed as untreated controls. We will continue recruitment until we have randomized a total of 146 cardiac transplant recipients. We will perform bone densitometry at randomization (unless performed within the previous month) and at 6 and 12 months. We will obtain radiographs (x-rays) at randomization and will repeat them at 12 months to detect undiagnosed vertebral fractures.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac transplantation

Exclusion Criteria:

* Active peptic ulcer disease, gastrectomy, inflammatory bowel disease, malignancy, Paget's disease of bone, osteogenesis imperfecta, multiple myeloma, primary hyperparathyroidism, rheumatoid arthritis, Cushing's syndrome, or thyrotoxicosis
* Suppressive doses of thyroid hormone, anticonvulsant drugs, past bisphosphonate therapy, current calcitonin therapy, or fluoride therapy
* Cirrhosis, inflammatory liver disease, or nephrolithiasis
* Serum creatinine > 2.5 mg/dl

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 1997-09; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shane, MD, Principal Investigator — Columbia University Department of Medicine
Locations (2):
- United States (2):
  - Columbai University Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York

REFERENCES:
- [Background] Shane E, Addesso V, Namerow PB, McMahon DJ, Lo SH, Staron RB, Zucker M, Pardi S, Maybaum S, Mancini D. Alendronate versus calcitriol for the prevention of bone loss after cardiac transplantation. N Engl J Med. 2004 Feb 19;350(8):767-76. doi: 10.1056/NEJMoa035617. PMID 14973216